CLINICAL TRIAL: NCT06519916
Title: Does a Gluten-free Diet Change the Mental Performance? A Comparative Study of Cognitive Function Among Children With Coeliac Disease and Healthy Controls
Brief Title: Mental Perfomance in Patients With Coeliac Disease
Status: Completed | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01095
Record Dates: First submitted 2024-05-28; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Celiac Disease in Children; Gluten Allergy
Keywords: mental performance; gluten-free diet; microbiome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with CD: Patients with CD, who have been diagnosed according to the Guidelines for diagnosing CD of the European Society for Paediatric Gastroenterology, Hepatology and Nutrition and stick strictly to a gluten-free diet (transglutaminase negative, at least for a year)
  Interventions: Behavioral: Assessment of mental performance
- Healthy control group: Age-and-sex-matched healthy control. Exclusion criteria for healthy controls were chronic diseases, regular medication intake, food allergies or specific diets.
  Interventions: Behavioral: Assessment of mental performance

INTERVENTIONS:
Behavioral: Assessment of mental performance — There was no intervention, the mental performance was assessed

SUMMARY:
Coeliac disease (CD) is an immune-mediated systemic disorder triggered by gluten in genetically predisposed patients. The only available treatment is a strict life long gluten-free diet (GFD), which has been linked to a reduced quality of life (QOL) and causes alterations in the gastrointestinal microbiome. Abnormal compositions of the microbiome are now recognized as factors in the pathogenesis of neuropsychological disorders via gut-brain-axis. The aim of this study was to assess the QOL and the mental performance of children and teenagers with CD and compare it to healthy controls (HC).

Methods: Children between the ages of 6 and 18 years with CD and age-and-sex-matched healthy controls (HC) filled in a questionnaire to assess QOL and performed the Flanker task, a standardized test to assess cognitive performance.

DETAILED DESCRIPTION:
Between July 2020 and August 2021, all children aged between 6 and 18 years, under the care of the University Children's hospital of Basel and the Children's hospital of Aarau, Switzerland, diagnosed with CD according to the Guidelines for diagnosing CD of the European Society for Paediatric Gastroenterology, Hepatology and Nutrition, were informed about the study. Further inclusion criteria were a strict adherence to the diet, defined as a negative transglutaminase for at least one year before participation in the study. Exclusion criteria comprised a diagnosis made less than a year ago, the presence of other chronic diseases, including food allergies, and the intake of regular medication. CD patients and their parents were informed about the study during the regular appointment for a clinical and serological check-up. After obtaining their consent, patients received another appointment to participate in the study.

For every CD-patient an age-and-sex-matched healthy control was recruited. Exclusion criteria for healthy controls were chronic diseases, regular medication intake, food allergies or specific diets.

Firstly, all participants were asked to fill in the questionnaire to examine the QOL. 'Kidscreen52' was used, a standardized questionnaire containing 52 questions, developed to assess the subjective health and the psychological, mental, and social well-being of children and adolescents covering ten important aspects of life (physical well-being, psychological well-being, moods & emotions, self-perception, autonomy, parent relation & home life, financial resources, peers & social support, school environment, bullying). The answers to all questions were converted into numbers from one to five. In most subgroups, a higher number indicates a more positive answer, except for 'self-perception' (questions are like: 'do you doubt your appearance' etc.) and 'bullying', where a lower number indicates also less exposure to bullying. Participants were also asked to fill in the ISI (insomnia severety index), a 7-item self-report standardized questionnaire assessing the nature, severity, and impact of insomnia.

Participants completed a computerized Flanker task to assess cognitive performance. In this cognitive task, the target was flanked by non-target stimuli, which correspond either to the same directional response as the target (congruent flankers) or to the opposite response (incongruent flankers). In our child-friendly variant, participants were presented with five fish in a row and were asked to press the correct button according to the orientation of the target (central fish). Participants were instructed to respond as accurately and as quickly as possible. The two different conditions were presented with equal probability. Visual stimuli were shown for 200 ms against a black background, followed by a blank inter-trial period of random length between 900 and 1300 ms. Participants completed one practice block and two test blocks with 40 trials each. Flanker task is a reliable, well-recognized neuropsychological test for assessing executive function . Mean reaction times (on response-correct trials) and accuracy rates were calculated for congruent and incongruent trials.

To have consistency, the interviews and instructions for Flanker task were conducted by the same three students. Uncomplete patient data sets were excluded.

ELIGIBILITY:
Inclusion Criteria:

* CD diagnosed according to European guidelines (ESPGHAN)
* only patients, who stick to a strict glutenfree diet (measured by transglutaminase for at least a year before participation in the study)

Exclusion Criteria: - any other chronic disease

-

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed with CD according to the Guidelines for diagnosing CD of the European Society for Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN), were informed about the study. Further inclusion criteria were a strict adherence to the diet, defined as a negative transglutaminase for at least one year before participation in the study
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Mental performance | cross-sectional
  The performance of the Flanker -Test was compared. Flanker-Test is a standardised test to assess mental performance. All participants performed this Flanker-Test (Computer Test) and afterwards the quality of life (see below ) was assessed. There was no follow-up, in this study participants with Coeliac disease and healthy controls only performed the Flanker-Test and the assessment of Quality of life (qol)and both groups were compared to each other. In other words, it is a snapshot, as the Flanker test and the quality of life survey were carried out on the same day.

SECONDARY OUTCOMES:
Quality of life (qol) | cross-sectional
  The outcome of qol was compared. To assess the quality of life, all participants had to fill in the questionnaire (Kidscreen-52) at the same time, than the Flanker-Test. All tests were performed within one year. Both tests were compared between the patients with Coeliac disease and the healthy control group. In other words, it is a snapshot, as the Flanker test and the quality of life survey were carried out on the same day.
  For the qol, the higher the score, the higher the qol

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Legeret, Principal Investigator — University Children's Hospital Basel
Locations (1):
- University Children's HOspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No